CLINICAL TRIAL: NCT02895971
Title: Incidence of Venous Thromboembolism and Professional Practices in Brest Area
Acronym: EPIGETBO III
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: EPIGETBO III (RB 12.157)
Record Dates: First submitted 2016-08-29; First posted 2016-09-12 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism; professional Practices
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study estimate VTE incidence. Investigators prospectively record all cases of symptomatic pulmonary embolism (PE) and deep vein thrombosis (DVT) of the lower limbs diagnosed between March 1, 2013 and February 28, 2014 in hospitals and in the community.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic pulmonary embolism (PE) and deep vein thrombosis (DVT) diagnosis confirmed
* Patient living in Brest area from time of diagnosis

Exclusion Criteria:

* invalid diagnosis
* asymptomatic event
* Main residence patient out of Brest area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with venous thromboembolism
Sampling Method: Probability Sample
Enrollment: 1416 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Gathering information about potential factors predisposing Thromboembolic disease and treatments undertaken. | two years after VTE
  After two years, all medication given to the patient to treat his initial VTE will be recorded, as well as the ongoing of thromboembolic disease

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France